CLINICAL TRIAL: NCT02290652
Title: Development and Validation of a Sexual Function Questionnaire for Female Patients Undergoing Total Hip Replacement
Brief Title: Sexual Function Questionnaire Total Hip Replacement
Status: Withdrawn | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 12/SC/0296
Record Dates: First submitted 2014-11-03; First posted 2014-11-14 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Arthritis
Keywords: Sexual function in Orthopaedic patients
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Prospective: Prospective - Factors affecting sexual function pre-THR
  Interventions: Other: Prospective - Factors affecting sexual function pre-THR
- Retrospective: Retrospective- Factors affecting sexual function post-THR
  Interventions: Other: Retrospective- Factors affecting sexual function post-THR

INTERVENTIONS:
Other: Prospective - Factors affecting sexual function pre-THR — A prospective assessment of factors affecting sexual function in patients whom are awaiting a total hip replacement.
  Patients will carry out a prospective 23 question questionnaire: 'Arthroplasty & Sexual Function Questionnaire (ASFQ) - Pre-operative' with validated questionnaire Female Sexual Function Index (FSFI), before their operation.
  Then at 6 months and 12 months post-operatively they will fill out a retrospective 30 question questionnaire: 'Arthroplasty & Sexual Function Questionnaire (ASFQ) - Post-operative', again with FSFI.
  Groups: Prospective
Other: Retrospective- Factors affecting sexual function post-THR — A retrospective assessment of factors affecting sexual function in patients whom have undergone a total hip replacement (THR) in the preceding year.
  Patients will carry out a retrospective 30 question questionnaire: 'Arthroplasty & Sexual Function Questionnaire (ASFQ) - Post-operative' with validated questionnaire Female Sexual Function Index (FSFI), at 6 months and/or 12 months (wherever possible).
  Maximum retrospective collection of data 12 months.
  Groups: Retrospective

SUMMARY:
* Non-commercial trial
* 2 Centres involved: University Hospital Southampton and Spire Southampton
* Expected number of eligible participants available per year: 100, (95% expected to agree to participation)
* The study will recruit prospectively female patients aged 18 - 65 years undergoing THR. A retrospective series of similar patients who have had a hip replacement will also be recruited.
* This is a research project that will run over 2 years. Data from 200 patients will be collected and analysed:

Retrospective 30 question questionnaire: 'Arthroplasty & Sexual Function Questionnaire (ASFQ) - Post-operative' Version 1.3 11/07/14

Prospective 23 question questionnaire: 'Arthroplasty & Sexual Function Questionnaire (ASFQ) - Pre-operative' Version 1.3 11/07/14

This project is significant in exploring an area of Orthopaedic medicine that has been little discussed in the literature. Preliminary results of our questionnaires have already revealed patients have a great desire to know how hip replacement will affect sexual function. Components of the questionnaire look at details such as: reasonable time frames for returning to sexual activity, positions that may be undesirable following replacement and which may lead to dislocation, concurrent use of analgesia and psychosexual aspects of total hip replacement surgery. The ultimate objective is to provide patients with detailed information about what to expect after hip replacement surgery.

DETAILED DESCRIPTION:
Prospective

Patients will be recruited from clinics at University Hospital Southampton and Spire Southampton Hospital. If they agree in principle to participate they will be provided with the Patient Information Sheet (PIS) and consent forms. Having completed the consent forms (one for participant to keep and one for the site file) participants are assigned an alphanumeric study number, which will be written at the top of all questionnaires and research paperwork completed. A form detailing demographic information will be filled out on recruitment to provide data for comparative quantitative analysis.

Prior to their operation, whether in hospital or by post (patient preference), they will complete a pre-operative ASFQ and FSFI questionnaire. These will be returned to the research team either in person (if completed by an inpatient) or returned in a pre-stamped addressed envelope. Copies of the National Joint Registry (NJR) data and PROMs will also be made and kept for evaluation alongside the questionnaire data. Patients will then complete the post-operative questionnaires and FSFI validated questionnaire at 6 and 12 months after their surgery. Questionnaires will be distributed to the patients in clinic at 6 months and sent to their home address at 12 months post-operatively (returned with stamped and addressed envelope).

Retrospective

Potential participant will be highlighted from previous inpatient list of patients eligible for participation. These patients will be contacted via telephone by a Good Clinical Practice (GCP) trained member of the research team member and invited to participate in the trial. If keen a PIS will be sent out to the patient's home address. The research team member will then follow-up with a phone-call to gain implied consent and complete an additional form detailing demographic information (the same information as the prospective cohort). The post-operative questionnaire, FSFI questionnaire and consent forms (one for participant to keep and one for the site file) with a stamped address envelope, will then be sent out to the participant to complete. Once documents are completed they will be returned to the research team. Questionnaires will be sent out at 6 and 12 months post-op where possible. Maximum time retrospective recruitment will be 12 months. The patient's NJR and PROMs will also be accessed for evaluation alongside the questionnaire data.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Sexually active
* Heterosexual
* 18- 65 years undergoing THR (prospective) or having undergone THR surgery within the last year

Exclusion Criteria:

* Sexually inactive pre-operatively and wishing to remain sexually inactive post-operatively
* Unable to comprehend English and with capacity to consent and follow instruction
* Unable to sign and date the ethics committee approved consent documentation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All female patients aged over 18 that are listed for a total hip replacement at University Hospital Southampton NHS Foundation Trust and The Spire Hospital Southampton that fulfill the inclusion criteria will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Factors affecting sexual activity related to total hip replacement, as measured by the Arthroplasty & Sexual Function Questionnaire (ASFQ) | 2 years
  To determine those patient and implant factors that affect sexual activity after hip replacement surgery. The study data will be used to publish an evidence-based patient information booklet that will be a standard reference for patients and healthcare professionals.

SECONDARY OUTCOMES:
Factors affecting sexual activity related to other joint replacement surgery, as measured by the Arthroplasty & Sexual Function Questionnaire (ASFQ) | 2-5 years
  The study will be extended to collect data from patients with knee arthritis who undergo knee replacement surgery (partial and total), as well as the partners of patients with hip and knee replacements. The study will also be extended to patients who have pre-arthritic conditions such as femoro-acetabular impingement, who undergo arthroscopic procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna C D'Souza, BM BSc(Hons), Principal Investigator — Research Fellow, UHS NHS FT.
Locations (2):
- United Kingdom (2):
  - Spire Southampton Hospital, Southampton, Hampshire
  - University of Southampton NHS Foundation Trust, Southampton, Hampshire